CLINICAL TRIAL: NCT00575978
Title: Hydralazine as Demethylating Agent in Breast Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: IRB request
Sponsor: University of Arkansas (Other)
Responsible Party: Ahmed Safar, MD, University of Arkansas for Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2003-23
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Hydralazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydralazine (Experimental): The objective of this study is to determine the MTD for hydrazaline added to standard neoadjuvant chemotherapy for operable breast cancer. Four dose levels of hydrazalline are planned:
  Dose Level 1: 150 mg/d 50 mg PO TID Dose Level 2: 200 mg/d 50 mg PO QID Dose Level 3: 225 mg/d 75 mg PO TID
  Interventions: Drug: Hydralazine

INTERVENTIONS:
Drug: Hydralazine — Dose Level 1: 150 mg/d 50 mg PO TID Dose Level 2: 200 mg/d 50 mg PO QID Dose Level 3: 225 mg/d 75 mg PO TID

SUMMARY:
This study will be conducted as a phase I/II clinical trial. In addition to determining the maximum tolerated dose (MTD) of hydralazine, the phase I trial will be performed to identify unexpected toxicities that may occur when hydralazine is used in conjunction with neoadjuvant chemotherapy in normotensive women with breast cancer. Once the phase I trial is successfully completed, the phase II trial to evaluate the efficacy of hydralazine in producing a demethylation effect will begin.

DETAILED DESCRIPTION:
The objective of this study is to determine the MTD for hydrazaline added to standard neoadjuvant chemotherapy for operable breast cancer. Four dose levels of hydrazalline are planned:

Dose Level 1: 150 mg/d 50 mg PO TID Dose Level 2: 200 mg/d 50 mg PO QID Dose Level 3: 225 mg/d 75 mg PO TID

Patients will be treated in cohorts of 3 and no patient may be treated at more that one dose level. Additional cohorts may not be initiated until toxicity has been fully evaluated in the current cohort of patients. The MTD is exceeded when a dose level produces a dose limiting toxicity (DLT) in at least two of the three patients in a cohort. Dose escalation will proceed by increasing the dose according to the following table.

Number of Events/Number in Cohort Action 0/3 Proceed to next dose level 1/3 Accrue 3 more patients at the same dose 1/3 + 0/3 Proceed to next dose level 1/3 + 1/3 Stop: Previous dose level is MTD 1/3 + 2/3 Stop: Previous dose level is MTD 1/3 + 3/3 Stop: Previous dose level is MTD 2/3 Stop: Previous dose level is MTD 3/3 Stop: Previous dose level is MTD

If the MTD has been exceeded by dose escalation and only one cohort with no observed toxicities was tested at the previous dose level, an additional cohort of 3 patients will be tested at the previous dose level. Thus, six patients must be treated at the dose declared the MTD. In the unlikely event that 150 mg/day of hydralazine, the starting dose, produces two or more DLTs, the daily dose of hydralazine will be reduced by 50mg to100 mg/day. If two or more toxicities are observed at this reduced dose level, the study will be stopped and the phase II study will not be performed.

This phase I study will require between 9 to 24 patients. The cohort of six patients treated at the MTD will be used in the subsequent phase II trial.

Definition of Dose Limiting Toxicities

Because the study drug is not a cytotoxic agent, is being "added" to a toxic chemotherapy regimen in women likely to be normotensive, and because the drug has been evaluated in the cardiovascular literature with maximum clinical doses at 300 mg/d, we made the following decisions that deviate from classic "cytotoxic" agent schemes. The deviations are as follows:

* Dose escalation beyond the "CLINNICALLY MAXIMAL" dose of 250 mg/d are not planned, and
* The definition of a DLT will not adhere to the NCI CTC - designed for cytotoxic agents, but will rather be simply the tolerability of the drug by the patient as documented in the protocol and reproduced below:

  1. Symptomatic hypotension,
  2. Blood pressure recording of < 90 mmHg systolic, or <55 mgHg diastolic,
  3. Other side effects deemed unacceptable either to the patient or the treating physician, and
  4. Patient request/refusal to continue on study.

Patients having to go off the drug will be considered as DLT events.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the breast cancer service for diagnostic evaluation for "breast growth" will be candidates to participate in this study. Patients with history of elevated blood pressure and who are already on anti-hypertensives would be ideal candidates for this project. In such situation, hydralazine will replace other anti-hypertensives. There is no age limit for this study. Inclusion criteria are as follows:

  1. Operable "invasive" breast cancer
  2. Signed informed consent
  3. Baseline blood pressure OFF antihypertensives > 110/60 mmHg

Exclusion Criteria:

1. Pre-existing hypotension
2. Pre-existing liver disease (liver function tests > 2x upper limits of normal ULM).
3. Pre-existing kidney (serum creatinine > 2 mg/dl).
4. Medical necessity to remain on beta-blockers that cannot be met by other agents.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-06; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To explore the potency of a clinical tolerable dose of hydralazine as a demethylating agent as indicated.

SECONDARY OUTCOMES:
1. Reversal of promoter methylation of eight Tumor Suppressor Genes (TSGs) reported as candidates for epigenetic silencing in breast cancer using Methylation-Specific

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Safar, MD, Principal Investigator — University of Arkansas